CLINICAL TRIAL: NCT04008446
Title: Effect of Vitamin B12 on the Development of Sepsis, in Culture Positive Patients : an Observational Study.
Brief Title: Effect of Vitamin B12 on the Development of Sepsis, in Culture Positive Patients
Acronym: Vit B12
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-00702
Record Dates: First submitted 2019-06-17; First posted 2019-07-05 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Bacteremia
MeSH Terms: conditions — Bacteremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bloodsample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an prospective observational study assessing the effect of vitamin B12 on the odds of developing sepsis in patients with infection confirmed by a positive culture result.

The hypothesis is that patients with infection confirmed by positive cultures who develop sepsis have lower vitamin B12 levels than patients infection, confirmed by positive cultures, who do not develop sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old)
* Infection, confirmed by a positive culture result
* Signed informed consent.

Exclusion Criteria:

* Pregnancy and/or breast feeding
* Inability to follow the procedures of the study, due to language problems, psychological disorders, social conditions or dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present to the ED with suspicion of infection, and for whom microbiological cultures are indicated,can to be enrolled into the study
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Holotranscobalamin (HTC) levels | 6 days
  HTC levels in patients with infection and sepsis compared to patients with infection without sepsis.

SECONDARY OUTCOMES:
Vitamin B12 levels | 6 days
  Levels of vitamin B12 in patients with infection and sepsis compared to patients with infection without sepsis
Methylmalonic acid (MMA) levels | 6 days
  Levels of ethylmalonic acid (MMA) in patients with infection and sepsis compared to patients with infection without sepsis

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pregernig A, Held U, Schlapfer M, Beck-Schimmer B. Vitamin B12 status and the risk of developing sepsis in patients with bacterial infection: a prospective observational cohort study. BMC Med. 2024 Aug 13;22(1):330. doi: 10.1186/s12916-024-03552-3. PMID 39134986